CLINICAL TRIAL: NCT00274079
Title: A Randomised, Double-blind, Parallel Group, 12 Week Study, Comparing the Effect of Once Daily Tiotropium Lactose Capsule With Placebo in Patients With Chronic Obstructive Pulmonary Disease (COPD), naïve to Anticholinergic Agents in Addition to Receiving Their Usual COPD Care
Brief Title: SPIRIVA in Ususal Care
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.276
Record Dates: First submitted 2006-01-09; First posted 2006-01-10 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

INTERVENTIONS:
Drug: SPIRIVA

SUMMARY:
The objective of the study is to determine the effect on lung function when either SPIRIVA once daily or placebo once daily is added to the usual therapy (care) of COPD patients naïve to anticholinergic agents managed in primary care. Previous studies have been in both hospital in and outpatients, with washout of some respiratory medications, this is the first study to be conducted in General Practice, the drug's anticipated environment.

Data from this study, including the adverse event monitoring, and post study findings on physical examination, will be used to extend the safety database. Health Resource Utilisation (HRU) data will be recorded to be use with data from other sources for economic analysis of COPD treatment.

DETAILED DESCRIPTION:
Anticholinergic drugs are currently indicated for all severities of COPD, due to the dominance of cholinergic tone in the pathological process of the disease. SPIRIVA is a new long acting anticholinergic, which has showed the benefits of improved lung function, dyspnoea, health status and less exacerbations compared to ipratropium, salmeterol and placebo in secondary care (hospital setting). The study will determine if the same effect is seen on the on lung function and dyspnoea when either SPIRIVA or placebo is added to the usual therapy /care of COPD patients naïve to anticholinergic agents managed in primary care.

The one year placebo and active controlled studies have confirmed efficacy and safety. No evidence of tolerance to the bronchodilator effects of tiotropium has been seen. Consistent improvements of health outcomes were also demonstrated. In the one-year studies, statistically significantly fewer patients in the tiotropium groups experienced exacerbations, or were hospitalised for exacerbations. Additionally, time to first exacerbation was increased. This suggests that moderate and severe exacerbations are reduced in-patients treated with tiotropium. The mechanism underlying this is not known, but may be associated with sustained airway opening.

The study will involve five visits to the GP surgery over a period of 14 weeks. Patient will attend for an initial visit to have the study information given to them and obtain their written consent. At the subsequent screening visit a physical examination including ECG together with an assessment of lung function will be performed. Once eligibility to the study is confirmed, and after completion of a 14 day 'run-in' period, patients will start treatment with a daily inhalation from the HandiHaler device of either SPIRIVA or placebo, this in addition to their usual COPD therapy.

Throughout the 12 week treatment period, patients will be required to inhale their study treatment medication (each morning) and complete a diary card. Patients will be required to return to the surgery after 2 and 6 weeks, with the final visit at 12 weeks for lung function testing, assessment of symptoms using the Oxygen Cost Diagram (OCD), Health Resources Utilisation (HRU) and any adverse events. On completion of the 12 week treatment period, a full physical examination will be repeated. Adverse event monitoring including COPD exacerbations will take place throughout the study.

Study Hypothesis:

Based on previous studies on COPD patients who were not on long acting beta agonists (LABAs), the standard deviation (SD) for trough FEV1 was 215 ml and an effect of 130 ml was seen on mean trough FEV1 with tiotropium.

It is assumed that 20% of primary care managed COPD patients will be using LABAs as part of their usual care. The effect of tiotropium on mean trough FEV1 in the study population is expected to be lower than the 130 ml seen in previous studies. Placebo is not expected to have any effect on mean trough FEV1.

Assuming an SD of 235ml, a total of 348 patients (174 per group) is adequate to detect a difference of 100 ml in mean trough FEV1 response between treatments with at the least 95% power at the 2.5% level of significance (one-sided) using a two group t-test.

To be considered complete, a patient must complete all primary efficacy data for all study visits as specified in the protocol without violations of the protocol so significant as to obscure the response to treatment.

Comparison(s):

Usual care for COPD

ELIGIBILITY:
Inclusion Criteria:

* Prior to participation in the study all patients must sign and date an informed consent consistent with ICH-GCP guidelines.
* Male or female patients 40 years of age or older.
* Patients with a diagnosis of COPD according to BTS criteria..A stable disease state with airway obstruction of FEV1 between 30- 65% of predicted normal value and FEV1 /FVC<70% pre bronchodilators.
* Predicted normal values will be calculated according to ECCS:
* For height measured in metres

  * Males: FEV1 predicted (L) = 4.30 X (Ht in mts) - 0.029 X (Age in yrs) - 2.49
  * Females:FEV1 predicted (L) = 3.95 X (Ht in mts) - 0.025 X (Age in yrs) - 2.60
* For height measured in inches

  * Males: FEV1 predicted (L) = 4.30 X (Ht in inches/39.37) - 0.029 X (Age in yrs) - 2.49
  * Females:FEV1 predicted (L) = 3.95 X (Ht in inches/39.37) - 0.025 X (Age in yrs) - 2.60
* Maintained on a stable respiratory medication for 4 weeks prior to visit 1 (no changes in respiratory medication oral dosage).
* Currently taking salbutamol or terbutaline MDI or DPI.
* Patient must be able to inhale medication through the HandiHaler?
* Patients must be able to perform technically acceptable pulmonary function tests in accordance with ATS criteria and must be able to maintain records (Patient Daily Record) during the study period as required in the protocol.
* Patients must be current or ex-smokers with a smoking history of more than 10 pack years.
* Pack Years = Number of cigarettes/day 20 (Patients who have never smoked cigarettes must be excluded.)

NOTE: An exacerbation of COPD requiring treatment occurring within the four week period prior to screening visit 1 will mean that screening should be postponed for at least four weeks. Therefore, the patient should have duration of at least 4 weeks free of exacerbations.

Exclusion Criteria:

* Patients with significant diseases, other than COPD will be excluded. A significant disease is defined as a disease which in the opinion of the investigator may either put the patient at risk because of participation in the study or a disease which may influence the results of the study or the patient's ability to participate in the study.
* Patients who have taken inhaled anticholinergics in the previous 12 months. Patients that have been treated with inhaled anticholinergics (via nebuliser or metered dose inhaler) due to an exacerbation for a time period no longer than 7 days may be included.
* Patients with an upper respiratory tract infection or exacerbation of COPD requiring treatment in the four weeks prior to the screening visit (visit 1) or during the two-week run-in period.

Patients with a recent history (i.e., six months or less) of myocardial infarction.

* Any unstable or life threatening cardiac arrhythmia requiring intervention or a change in drug therapy within the last year.
* Patients with known active tuberculosis.
* Patients who have a history of thoracotomy with pulmonary resection or have planned lung transplantation or lung volume reduction surgery.
* Patients with a history of asthma, cystic fibrosis, bronchiectasis, interstitial lung disease or pulmonary thromboembolic disease.
* Patients who are being treated with antihistamines (H1 receptor antagonists) for asthma or excluded allergic conditions.
* Patients with a history of cancer in the last five years; Basal cell tumours or patients whose length of time in remission is greater than five years can be included.
* Patient with known hypersensitivity to atropine, and other anticholinergic drugs or lactose or any previous adverse reaction to anticholinergic drugs that resulted in withdrawal of the anticholinergic compound.
* Patients using oral corticosteroid medication at unstable doses (i.e. Patients have been on a stable dose for less than 6 weeks prior to randomisation) or at doses in excess of the equivalent of 10mg o

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 395
Dates: Start 2002-10; Primary Completion 2003-10 (Actual); Study Completion 2003-10

PRIMARY OUTCOMES:
Trough Forced Expiratory Volume in one second (FEV1) response determined at the end of the 12- week treatment period | week 12

SECONDARY OUTCOMES:
Trough FEV1 response after 2 and 6 weeks | week 2, week 6
Trough Forced Vital Capacity (FVC) response after 2, 6 and 12 weeks | week 2, week 6, week 12
Dyspnoea measured by the Oxygen Cost Diagram (OCD | week 12
Weekly mean number per day of occasions when Short Acting β2 Agonist (SABA) therapy was used | week 12
Percentage compliance with study medication as assessed by inhalation capsule counts | week 12
Adverse events | week 12
Seated pulse rate and blood pressure | week 12
Physical examination | week 12

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Boehringer Ingelheim Ltd./Bracknell
Locations (38):
- United Kingdom (38):
  - Foresterhill Healthcentre, Aberdeen
  - Boehringer Ingelheim Investigational Site, Airdrie
  - Boehringer Ingelheim Investigational Site, Atherstone
  - Boehringer Ingelheim Investigational Site, Barry
  - Boehringer Ingelheim Investigational Site, Bath
  - The Beehive Surgery, Bath, Bath
  - Boehringer Ingelheim Investigational Site, Bedworth
  - Boehringer Ingelheim Investigational Site, Bellshill
  - Boehringer Ingelheim Investigational Site, Bexhill-on-Sea
  - Health Centre, Biggar
  - Bradford Health Centre, Bradford Upon Avon
  - Pembroke Road Surgery, Bristol
  - Boehringer Ingelheim Investigational Site, Cardiff
  - Boehringer Ingelheim Investigational Site, Chapelhall
  - Boehringer Ingelheim Investigational Site, Coatbridge
  - Coatbridge Health Centre, Coatbridge
  - Boehringer Ingelheim Investigational Site, Corsham
  - Boehringer Ingelheim Investigational Site, Coventry
  - Boehringer Ingelheim Investigational Site, Doncaster
  - Boehringer Ingelheim Investigational Site, Garston
  - Boehringer Ingelheim Investigational Site, Glasgow
  - Boehringer Ingelheim Investigational Site, Glenboig
  - Princess Street Surgery, Gorseinon
  - Boehringer Ingelheim Investigational Site, Hamilton
  - Boehringer Ingelheim Investigational Site, Haverfordwest
  - Boehringer Ingelheim Investigational Site, Heywood
  - Boehringer Ingelheim Investigational Site, Holt
  - Boehringer Ingelheim Investigational Site, Kingswood
  - Boehringer Ingelheim Investigational Site, Leicester
  - Boehringer Ingelheim Investigational Site, Melksham
  - Boehringer Ingelheim Investigational Site, Plymouth
  - St Chads Surgery, Radstock
  - Boehringer Ingelheim Investigational Site, Royal Leamington Spa
  - Boehringer Ingelheim Investigational Site, Rutherglen
  - Boehringer Ingelheim Investigational Site, Sheffield
  - Boehringer Ingelheim Investigational Site, Soham
  - Boehringer Ingelheim Investigational Site, Wishaw
  - Boehringer Ingelheim Investigational Site, Woking

REFERENCES:
- [Derived] Freeman D, Lee A, Price D. Efficacy and safety of tiotropium in COPD patients in primary care--the SPiRiva Usual CarE (SPRUCE) study. Respir Res. 2007 Jul 2;8(1):45. doi: 10.1186/1465-9921-8-45. PMID 17605774